CLINICAL TRIAL: NCT02828865
Title: A Prospective Clinical Trial Using Irreversible Electroporation for the Treatment of Liver Cancers
Brief Title: A Clinical Trial Using Irreversible Electroporation for the Treatment of Liver Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201210007DIC
Record Dates: First submitted 2016-06-27; First posted 2016-07-12 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Metastatic Liver Cancers
Keywords: Hepatocellular Carcinoma; irreversible electroporation; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Electroporation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irreversible electroporation (IRE) (Experimental): irreversible electroporation (IRE) (AngioDynamics, NY) To use 2 to 6 unipolar electrodes of IRE in a predetermined grid pattern. 90 pulses of 2,000 - 3,000 V were applied with a pulse generator (AngioDynamics, NY) across the gap between the electrodes for 100 microseconds (0.1 msec) per each ablation.
  Interventions: Device: Irreversible Electroporation (IRE) System

INTERVENTIONS:
Device: Irreversible Electroporation (IRE) System

SUMMARY:
Liver cancer including primary hepatocellular carcinoma (HCC) and metastatic liver cancers is one the most common malignancies in the world. Over 10000 new cases per year are diagnosed in Taiwan. Despite the many treatment options, the prognosis of HCC remains dismal. More than 8000 people died of this cancer every year in Taiwan. A majority (70% to 85%) of patients present with advanced or unresectable disease. In contrast, small liver cancers can be cured with an appreciable frequency. Five-year disease-free survival exceeding 50% has been reported for surgical resection, and for the inoperable patients who do not have vascular invasion or extrahepatic spread. Radiofrequency ablation (RFA) is recommended as an alternative curative therapy. However, the main drawback of RFA is its limitation to tumor size and location. The tumors larger than 5 cm in diameter or located adjacent to vessels, could not be ablated completely sometimes.

DETAILED DESCRIPTION:
Irreversible electroporation (IRE), developed and manufactured by AngioDynamics US Ltd, can ablate tumor by fenestrating the cancer cell membrane by electric pulse. The anti-tumor effect does not result from thermotherapy, so is also not diminished by adjacent vessels. Several pre-clinical studies have already demonstrated IRE is a safe and effective treatment for live cancers. The system has been approved as safe by the European Union (EU) in 2008 and received Food and Drug Administration (FDA) approval in 2010. However, there are still few experiences in using IRE for tumor ablation in Taiwan. In this study, the investigators will perform IRE for 40 inoperable patients with liver cancers adjacent to vessels who are suitable to receive radiofrequency ablation (RFA) in the investigators hospital. The investigators will evaluate the potential side effect and ablate effect of tumors by abdominal computed tomography (CT) or magnetic resonance imaging (MRI), and the investigators will also follow-up this patients for 2 years to evaluate the overall survival and local recurrence rate. The investigators will appraisal the clinical feasibility and advantage of the system by this study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. The diagnosis of hepatocellular carcinoma (HCC) or metastatic liver cancers with pathologic proven, and the diagnosis of HCC will be made by pathology / cytology or according to the American Association for the Study of Liver Diseases (AASLD) (2010) diagnostic criteria. In brief, Nodules larger than 1 cm found on ultrasound screening of a cirrhotic liver should be investigated further with either tri-phase multidetector computed tomography (CT) scan or dynamic contrast enhanced magnetic resonance imaging (MRI). If the appearances are typical of HCC (i.e., hypervascular in the arterial phase with washout in the portal venous or delayed phase), the lesion should be treated as HCC. If the findings are not characteristic or the vascular profile is not typical, a second contrast enhanced study with the other imaging modality should be performed, or the lesion should be biopsied. Biopsies of small lesions should be evaluated by expert pathologists. Tissue that is not clearly HCC should be stained with all the available markers including cluster of differentiation 34 (CD34), cytokeratin 7 (CK7), glypican 3, heat shock protein 70 (HSP70), and glutamine synthetase to improve diagnostic accuracy.
2. Unsuitable for surgical resection but local ablation is indicated, however, the distance between tumour and vessels is smaller than 5 mm.
3. Have at least one, but less than or equal to 3 tumors,
4. Each tumor must be ≤ 5 cm in diameter,
5. Child-Pugh class A-B,
6. Eastern Cooperative Oncology Group (ECOG) score of 0-1,
7. American Society of Anaesthesiologists (ASA) score ≤ 3,
8. Adequate bone marrow, liver and renal function. Platelet count ≥ 100 K/Μl. Total bilirubin ≦ 2 mg/dL. alanine transaminase (ALT) and aspartate transaminase (AST) < 5 x upper limit of normal. prothrombin time (PT)- international normalized ratio (INR) ≦ 2.0. Serum creatinine ≦ 1.5 x upper limit of normal
9. Prior Informed Consent Form
10. Life expectancy of at least 3 months.
11. The disease status is not suitable to receive surgical resection, percutaneous alcohol injection, transarterial chemoembolization or other standard treatment.

Exclusion Criteria:

Patients presenting with any of the following will not be enrolled into this study:

1. History of cardiac disease:

1. Congestive heart failure >New York Heart Association (NYHA) class 2
2. Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed)
3. Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 3.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker
4. Uncontrolled hypertension 2. Any active metal implanted device (eg Pacemaker), 3. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception, 4. Received treatment with an investigational agent/ procedure within 30 days prior to treatment with the IRE System, 5. Known history of HIV infection 6. Concurrent extrahepatic cancer

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12-18 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Tumor response | 1 month after treatment
  Tumor response, according to modified RECIST criteria, will be evaluated by abdominal computed tomography (CT) or magnetic resonance imaging (MRI) 1 month after treatment.

SECONDARY OUTCOMES:
Change of Eastern Cooperative Oncology Group (ECOG) evaluation | one to two years
  Complete an Eastern Cooperative Oncology Group (ECOG) evaluation
Change of vital signs | one to two years
  Measure vital signs including temperature, respiratory rate, blood pressure, and heart rate.
Physical examination | one to two years
  Conduct a physical examination.
Clinical laboratory assessments | one to two years
  Collect blood samples for Clinical laboratory assessments, including hematology, A-fetoprotein (AFP) (for hepatocellular carcinoma (HCC)) / carcinoembryonic antigen (CEA) (for adenocarcinoma) and chemistry evaluations.
Urinalysis | one to two years
  Collect urine sample for a routine urinalysis.
Conduct CT or MR scans for tumour response evaluation | one to two years
  Subjects will still be followed-up in the event of disease progression in order to document local recurrence, a secondary endpoint.
Review concomitant medications | one to two years
  Use of medications will be reviewed and recorded.
Assess for presence of adverse events | one to two years
  An adverse event assessment will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No